CLINICAL TRIAL: NCT03977415
Title: Interstitial Lung Disease in Early Rheumatoid Arthritis
Acronym: ILD-Early RA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: HS-3140
Record Dates: First submitted 2018-07-26; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Rheumatoid Arthritis; Interstitial Lung Disease
Keywords: Interstitial Lung Disease; ILD; Pulmonary Fibrosis; Rheumatoid Arthritis; RA; Rheumatology
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum biomarker and cell collection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA with no ILD: Subjects diagnosed with RA less then 2 years and without a diagnosis of ILD, will complete 5 in-person study visits. Visits will be performed every 6 months for 18 months.
  Study Assessments Include:
  1. Medical history and Physical exams
  2. Quality of Life Questionnaires
  3. Collection of Sputum and Blood
  4. Radiology (HRCT)
  5. Lung Function Test
- RA with ILD: Patients diagnosed with RA less than 2 years, and clinically diagnosed with interstitial lung disease (ILD), will complete 5 in-person study visits. Visits will be performed every 6 months for 18 months.
  Study Assessments Include:
  1. Medical history and Physical exams
  2. Quality of Life Questionnaires
  3. Collection of Sputum and Blood
  4. Radiology (HRCT)
  5. Lung Function Test
  6. Spirometry

SUMMARY:
The purpose of this study is to determine how interstitial lung disease can be predicted over time in early rheumatoid arthritis. The investigators will study blood and phlegm samples from participants, along with quality of life questionnaires to determine if and how the presence of ILD may impact the participants quality of life over time.

DETAILED DESCRIPTION:
Participation involves 5 study visits over an 18 month timeframe. During each of these visits, a recent medical history and physical exam will take place, blood and phlegm will be collected, quality of life questionnaires will be administered, and a CT-scan of the chest and pulmonary function testing may be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 90 years
2. Diagnosis of "early RA" with or without ILD as defined by ACR/EULAR 2010 criteria and confirmed by a member of the ILD or Rheumatology programs at National Jewish Health (NJH)
3. Able to read, speak, and understand English
4. Able and willing to perform all study related tasks, including returning to NJH every 6 months for an 18 month period of time

Exclusion Criteria:

1. Subjects who do not meet all inclusion criteria
2. Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are selected for participation in the study because they have an active diagnosis of rheumatoid arthritis and are at risk fro the development of lung disease.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in anti-CCP antibody test to identify the presence or development of RA in patients with or without ILD | 18 months
Change in lung antigen targets in RA-ILD using induced sputum | 18 months
Change from baseline for Leicester Cough questionnaire-Acute (LCQ_Acute) | 18 months
Change from baseline for Short Form (SF_36) questionnaire | 18 months
Change from baseline for UCSD Medical Center Pulmonary Rehabilitations Program Shortness-of-Breath questionnaire | 18 months
Change from baseline for Multi-Dimensional Health Assessment questionnaire (MDHAQ) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Solomon, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States